CLINICAL TRIAL: NCT02565693
Title: Apixaban Versus Antiplatelet Drugs or no Antithrombotic Drugs After Anticoagulation-associated Intracerebral Haemorrhage in Patients With Atrial Fibrillation: A Randomised Phase II Clinical Trial
Brief Title: Apixaban After Anticoagulation-associated Intracerebral Haemorrhage in Patients With Atrial Fibrillation
Acronym: APACHE-AF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Heart Foundation (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, H. Bart van der Worp, Co-Coordinating Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL47761.041.14; 2014-000112-33 (EudraCT Number); NTR4526 (Registry Identifier: Nederlands Trialregister); U1111-1154-5474 (Registry Identifier: WHO Universal Trial Number)
Record Dates: First submitted 2015-08-27; First posted 2015-10-01 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Hemorrhage; Atrial Fibrillation
MeSH Terms: conditions — Cerebral Hemorrhage; Atrial Fibrillation | interventions — apixaban; Aspirin; carbaspirin calcium; Clopidogrel; Dipyridamole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban (Experimental): Apixaban: oral, 5 mg twice daily. If two of the three following criteria are met, the dose will be reduced to 2.5 mg twice daily:
  * Age ≥ 80 years
  * Body weight ≤ 60 kg
  * Serum creatinine ≥ 133 μmol. Additionally, if the creatinin clearance is below 30 ml per minute, the dose will be reduced to 2.5 mg twice daily.
  Interventions: Drug: Apixaban
- Avoiding oral anticoagulants (Other): The following treatment regimens are allowed in the comparator arm:
  - No antithrombotic treatment
  or:
  * Acetylsalicylic acid 80 mg once daily
  * Carbasalate calcium 100 mg once daily
  * Clopidogrel 75 mg once daily
  * Acetylsalicylic acid 80 mg once daily and dipyridamole 200 mg twice daily
  * Carbasalate calcium 100 mg once daily and dipyridamole 200 mg twice daily
  Interventions: Drug: Aspirin; Drug: Carbasalate calcium; Drug: Clopidogrel; Drug: Dipyridamole; Other: No antithrombotic treatment

INTERVENTIONS:
Drug: Apixaban
  Other Names: Eliquis
  Arms: Apixaban
Drug: Aspirin
  Other Names: Acetylsalicylic acid
  Arms: Avoiding oral anticoagulants
Drug: Carbasalate calcium
  Arms: Avoiding oral anticoagulants
Drug: Clopidogrel
  Arms: Avoiding oral anticoagulants
Drug: Dipyridamole
  Arms: Avoiding oral anticoagulants
Other: No antithrombotic treatment
  Arms: Avoiding oral anticoagulants

SUMMARY:
There is a marked lack of evidence on the optimal prevention of ischaemic stroke in patients with atrial fibrillation and a recent intracerebral haemorrhage (ICH) during treatment with oral anticoagulation. These patients are currently treated with vitamin K antagonists, DOACs, antiplatelet drugs, or no antithrombotic treatment, depending on personal and institutional preferences. Treatment with a direct oral anticoagulant like apixaban might be an attractive alternative in terms of a low risk of recurrent ICH, while at the same time being effective for the prevention of ischaemic stroke. This study aims to obtain reliable estimates of the rates of vascular death or non-fatal stroke in patients with atrial fibrillation and a recent anticoagulation-associated intracerebral haemorrhage who are treated with apixaban versus those who are treated with antiplatelet drugs or no antithrombotic drug at all.

This study has a multi-centre, phase II, randomised, open-label clinical trial with blinded outcome assessment design.

DETAILED DESCRIPTION:
Rationale: There is a marked lack of evidence on the optimal prevention of ischaemic stroke and other thrombo-embolic events in patients with non-valvular atrial fibrillation (AF) and a recent intracerebral haemorrhage (ICH) during treatment with oral anticoagulation. These patients are currently treated with oral anticoagulants, antiplatelet drugs, or no antithrombotic treatment, depending on personal and institutional preferences. Randomised trials in patients with AF but without ICH have convincingly shown that vitamin K antagonists (VKAs, such as warfarin) reduce the risk of ischaemic stroke and other thrombo-embolic events, but increase the risk of bleeding as compared to no anticoagulant therapy. In the ARISTOTLE trial, the direct oral anticoagulant (DOAC) apixaban was superior to warfarin in preventing stroke or systemic embolism, caused less bleeding, and resulted in lower mortality. In other trials, the other DOACs, rivaroxaban, edoxaban, and dabigatran had a similar benefit as compared with warfarin. DOACs have not been tested in patients with AF and a recent ICH. Apixaban is the only DOAC tested against aspirin in a large randomised trial, in which patients with AF who were treated with apixaban had a lower risk of stroke or systemic embolism than those treated with aspirin, whereas ICH rates were similar in both treatment groups. We hypothesize that in patients with AF who survived an anticoagulation-associated ICH, apixaban is an attractive alternative to antiplatelet drugs or no antithrombotic treatment at all in terms of a low risk of recurrent ICH, while at the same time being more effective for the prevention of ischaemic stroke.

Objective: 1) To obtain reliable estimates of the rates of vascular death or non-fatal stroke in patients with atrial fibrillation and a recent anticoagulation-associated intracerebral haemorrhage who are treated with apixaban versus those who are treated with an antiplatelet drug or no antithrombotic drugs. 2) To compare the rates of all-cause death, stroke, ischaemic stroke, ICH, other major haemorrhage, systemic embolism, and functional outcome between patients treated with apixaban and those who are treated with an antiplatelet drug or no antithrombotic drugs.

Study design: A randomised, open, multi-center clinical trial with masked outcome assessment.

Study population: 100 adults with a history of atrial fibrillation and a recent intracerebral haemorrhage during treatment with anticoagulation in whom clinical equipoise exists on the optimal stroke prevention therapy.

Intervention: Apixaban 5 mg twice daily versus antiplatelet therapy or no antithrombotic drugs.

Primary outcome: Vascular death or non-fatal stroke during follow-up. Time frame: We aim to include 100 patients in six years. All patients will be followed up for the duration of the study, but at least for six months.

ELIGIBILITY:
Inclusion Criteria:

* Intracerebral haemorrhage (including including isolated spontaneous intraventricular haemorrhage), documented with CT or MRI, during treatment with anticoagulation (VKA, any direct thrombin inhibitor, any factor Xa inhibitor, or (low molecular weight) heparin at a therapeutic dose).
* The haemorrhage has occurred between 7 and 90 days before randomization.
* Diagnosis of (paroxysmal) non-valvular AF, documented on electrocardiography.
* A CHA2DS2-VASc score ≥ 2.
* Score on the modified Rankin scale (mRS)≤4.
* Equipoise regarding the optimal medical treatment for the prevention of stroke.
* Age ≥ 18 years.
* Written informed consent by the patient or by a legal representative

Exclusion Criteria:

* Conditions other than atrial fibrillation for which the patient requires long-term anticoagulation
* A different clinical indication for the use of an antiplatelet drug even if treated with apixaban, such as clopidogrel for recent coronary stenting.
* Mechanical prosthetic heart valve (biological prosthetic heart valves are allowed) or rheumatic mitral valve disease.
* Serious bleeding event in the previous 6 months, except for intracerebral haemorrhage.
* High risk of bleeding (e.g., active peptic ulcer disease, a platelet count of <100,000.mL-1 or haemoglobin level of <6.2 mMol.L-1, ischaemic stroke in the previous 7 days (patients are eligible thereafter), documented haemorrhagic tendencies, or blood dyscrasias).
* Current alcohol or drug abuse.
* Life expectancy of less than 1 year.
* Severe renal insufficiency (a serum creatinine level of more than 221 μmol per liter or a calculated creatinine clearance of <15 ml per minute).
* Alanine aminotransferase or aspartate aminotransferase level greater than 2 times the upper limit of the normal range or a total bilirubin more than 1.5 times the upper limit of the normal range, unless a benign causative factor (e.g. Gilbert's syndrome) is known or identified.
* Allergy to apixaban.
* Use of strong cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp) inhibitors (e.g. systemic azole-antimycotics as ketoconazole or HIV protease inhibitors such as ritonavir).
* Pregnancy or breastfeeding.
* Women of childbearing potential: any woman who has begun menstruation and is not postmenopausal or otherwise permanently unable to conceive. A postmenopausal woman is defined as a woman who is over the age of 45 and has not had a menstrual period for at least 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who experience the combination of vascular death or non-fatal stroke (cerebral infarction, intracerebral haemorrhage, or subarachnoid haemorrhage) | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  Ischaemic stroke Clinical evidence of the sudden onset of an new neurological deficit, or an increase in an existing deficit, persisting for more than 24 hours, without evidence of a intracerebral haemorrhage on a CT or MRI scan or at post-mortem investigation.
  Intracerebral haemorrhage Clinical evidence of the sudden onset of a new neurological deficit, or an increase in an existing deficit, persisting for more than 24 hours, with a corresponding intracerebral haemorrhage on a CT or MR scan or at post-mortem investigation.
  Unclassified stroke Clinical evidence of the sudden onset of a new neurological deficit, or an increase in an existing deficit, persisting for more than 24 hours, without imaging or post-mortem investigations performed.
  Subarachnoid haemorrhage Subarachnoid haemorrhage (SAH) demonstrated by CT, lumbar puncture, or at post-mortem investigation.
  Vascular death See Outcome 2, Vascular death

SECONDARY OUTCOMES:
Number of patients who experience vascular death | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
Number of patients who experience death from any cause. | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  Vascular death Death from cerebral infarction; intracerebral, subarachnoid, epidural, or subdural haemorrhage; unclassified stroke; myocardial infarction; extracranial haemorrhage; or systemic embolism. Death should have been unlikely without the events mentioned above. Other events classifying as vascular death: fatal arterial or gastric bleeding, terminal heart failure, fatal pulmonary embolism, and sudden death, defined as death within one hour after onset of symptoms.
Number of patients who experience all stroke. | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  Ischaemic stroke Clinical evidence of the sudden onset of an new neurological deficit, or an increase in an existing deficit, persisting for more than 24 hours, without evidence of a intracerebral haemorrhage on a CT or MRI scan or at post-mortem investigation.
  Intracerebral haemorrhage Clinical evidence of the sudden onset of a new neurological deficit, or an increase in an existing deficit, persisting for more than 24 hours, with a corresponding intracerebral haemorrhage on a CT or MR scan or at post-mortem investigation.
  Unclassified stroke Clinical evidence of the sudden onset of a new neurological deficit, or an increase in an existing deficit, persisting for more than 24 hours, without imaging or post-mortem investigations performed.
  Subarachnoid haemorrhage Subarachnoid haemorrhage (SAH) demonstrated by CT, lumbar puncture, or at post-mortem investigation.
Number of patients who experience ischaemic stroke. | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  Clinical evidence of the sudden onset of an new neurological deficit, or an increase in an existing deficit, persisting for more than 24 hours, without evidence of a intracerebral haemorrhage on a CT or MRI scan or at post-mortem investigation.
Number of patients who experience intracerebral haemorrhage. | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  Clinical evidence of the sudden onset of a new neurological deficit, or an increase in an existing deficit, persisting for more than 24 hours, with a corresponding intracerebral haemorrhage on a CT or MR scan or at post-mortem investigation.
Number of patients who experience other major extracranial haemorrhage | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  Major extracranial bleeding will be defined using the ISTH criteria.55 1) Fatal bleeding, and/or 2) Symptomatic bleeding in a critical area or organ, such as intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or 3) Bleeding causing a fall in haemoglobin level of 1.24 mmol L-1 or more, or leading to transfusion of two or more units of whole blood or red cells.
  ￼￼￼
Number of patients who experience any intracranial haemorrhage other than ICH. | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  subdural haemorrhage: evidence of a subdural haematoma on a CT or MRI scan or at post-mortem investigations; epidural hematoma: evidence of an epidural haematoma on a CT or MRI scan or at post-mortem investigations.
Number of patients who experience systemic embolism. | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  The diagnosis of systemic embolism requires a clinical history consistent with an acute loss of blood flow to a peripheral artery (or arteries) supported by evidence of embolism from surgical specimens, post-mortem investigations, angiography, vascular imaging, or other objective testing.
Number of patients who experience myocardial infarction. | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  Detection of a rise and/or fall of cardiac biomarker values [preferably cardiac troponin] with at least 1 value above the 99th percentile upper reference limit and with at least 1 of the following:
  Symptoms of ischemia. New or presumed new significant ST-segment-T wave changes or new left bundle branch block. Development of pathological Q waves in the ECG. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality. Identification of intracoronary thrombus by angiography or autopsy.
  Cardiac death with symptoms suggestive of myocardial ischemia and presumed new ischemic ECG changes or new LBBB, but death occurred before cardiac biomarkers were obtained, or before cardiac biomarker values would be increased.
Number of patients who experience who experience a good functional outcome as assessed with the score on the modified Rankin Scale | Throughout the study. Patients will be followed up between 12 (minimum) and 72 (maximum) months.
  Van Swieten JC, Koudstaal PJ, Visser MC, Schouten HJ, van Gijn J. Interobserver agreement for the assessment of handicap in stroke patients. Stroke. 1988 May;19(5):604-7.

CONTACTS AND LOCATIONS:
Overall Officials: Catharina JM Klijn, MD PhD, Study Chair — Radboud University Medical Center; H Bart van der Worp, MD PhD, Study Chair — UMC Utrecht
Locations (16):
- Netherlands (16):
  - Amsterdam UMC, Amsterdam
  - OLVG, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Zuyderland Ziekenhuis, Heerlen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC, Rotterdam
  - Haaglanden MC, The Hague
  - Elisabeth-Tweesteden Ziekenhuis, Tilburg
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Schreuder FHBM, van Nieuwenhuizen KM, Hofmeijer J, Vermeer SE, Kerkhoff H, Zock E, Luijckx GJ, Messchendorp GP, van Tuijl J, Bienfait HP, Booij SJ, van den Wijngaard IR, Remmers MJM, Schreuder AHCML, Dippel DW, Staals J, Brouwers PJAM, Wermer MJH, Coutinho JM, Kwa VIH, van Gelder IC, Schutgens REG, Zweedijk B, Algra A, van Dalen JW, Jaap Kappelle L, Rinkel GJE, van der Worp HB, Klijn CJM; APACHE-AF Trial Investigators. Apixaban versus no anticoagulation after anticoagulation-associated intracerebral haemorrhage in patients with atrial fibrillation in the Netherlands (APACHE-AF): a randomised, open-label, phase 2 trial. Lancet Neurol. 2021 Nov;20(11):907-916. doi: 10.1016/S1474-4422(21)00298-2. PMID 34687635
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170